CLINICAL TRIAL: NCT03745105
Title: Comparative Evaluation of the Effect of a Prophylactic Intraligamentary Injection of Dexamethasone and Piroxicam on Postoperative Pain in Teeth With Symptomatic Irreversible Pulpitis: A Randomized Controlled Trial
Brief Title: Comparative Evaluation of the Effect of Prophylactic Intraligamentary Injection of Dexamethasone and Piroxicam on Postoperative Pain in Teeth With Symptomatic Irreversible Pulpitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Safwa Essam Mohammed Ahmed Abd el-glil, resident at faculty of dentistry cairo university, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEBD-CU-2018-11-01
Record Dates: First submitted 2018-11-13; First posted 2018-11-19 (Actual); Last update posted 2018-11-23 (Actual); Status verified 2018-11

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — dexamethasone 21-phosphate; Mepivacaine

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- dexamethasone (Experimental): Pretreatment intraligamentary injection of 0.4 mL of 8 mg/2 mL dexamethasone (Dexamethasone, AMRIYA pharmaceutical, Egypt)
  Interventions: Drug: Dexamethasone sodium phosphate
- piroxicam (Experimental): Pretreatment intraligamentary injection of 0.4 mL of 20 mg mL-1 piroxicam (Feldene, Pfizer, Egypt)
  Interventions: Drug: Piroxicam Injectable Solution
- Mepivacaine HCL (Active Comparator): Pretreatment Intraligamentary injection of 0.4 mL of Mepivacaine HCl 36 mg /1.8 ml + Levonordefrin HCl 0.108 mg/ 1.8 ml (Mepecaine - L, Alexandria Co.-Egypt)
  Interventions: Drug: Mepivacaine HCL

INTERVENTIONS:
Drug: Dexamethasone sodium phosphate — prophylactic intraligamentary supplemental injection of 0.4 ml of 8 mg/2 mL dexamethasone.
  Arms: dexamethasone
Drug: Piroxicam Injectable Solution — prophylactic intraligamentary supplemental injection of 0.4 mL of 20 mg mL-1 piroxicam
  Arms: piroxicam
Drug: Mepivacaine HCL — prophylactic intraligamentary supplemental injection 0.4 mL of Mepivacaine HCl 36 mg /1.8 ml + Levonordefrin HCl 0.108 mg/ 1.8 ml
  Arms: Mepivacaine HCL

SUMMARY:
the study is conducted to assess and compare the efficacy of local intraligamentary injection of glucocorticoids(dexamethasone) and NSAID(piroxicam) on reduction of postoperative pain in patients with symptomatic irreversible pulpitis.

ELIGIBILITY:
Inclusion Criteria:

1. Systemically healthy patient (ASA I or II).
2. Mandibular Posterior teeth with:

   * Preoperative sharp pain.
   * Absence of widening in the periodontal ligament (PDL).
   * Vital response of pulp tissue to cold pulp tester (ethyl chloride spray).

Exclusion Criteria:

1. Patients allergic to anesthetics, piroxicam (any other NSAIDs) or dexamethasone (other corticosteroids).
2. Pregnant or nursing females.
3. Patients having significant systemic disorder (ASA III or IV).
4. Hemostatic disorders or anti-coagulant therapy during the last month.
5. Consumption of opioid or non-opioid analgesics or corticosteroids during the last 12 hrs before treatment.
6. Retreatment cases.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2018-12-25 (Estimated); Primary Completion 2019-12-01 (Estimated); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
Post operative pain assessed with the Numerical Rating Pain Scale | up to 48 hours after root canal treatment (At 4,6,12,24 and 48 hours after root canal treatment ).
  Intensity of pain after endodontic treatment is recorded by the patient using a numerical rating scale(where 0= no pain ,1-3 =mild pain ,4-6= moderate pain and 7-9= severe pain )

SECONDARY OUTCOMES:
number of analgesics taken by the patient | Until 48 hours after endodontic treatment.
  Number of analgesic tablets taken by the patient after endodontic treatment.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mehrvarzfar P, Esnashari E, Salmanzadeh R, Fazlyab M, Fazlyab M. Effect of Dexamethasone Intraligamentary Injection on Post-Endodontic Pain in Patients with Symptomatic Irreversible Pulpitis: A Randomized Controlled Clinical Trial. Iran Endod J. 2016 Fall;11(4):261-266. doi: 10.22037/iej.2016.2. PMID 27790253
- [Background] Atbaei A, Mortazavi N. Prophylactic intraligamentary injection of piroxicam (feldene) for the management of post-endodontic pain in molar teeth with irreversible pulpitis. Aust Endod J. 2012 Apr;38(1):31-5. doi: 10.1111/j.1747-4477.2010.00274.x. Epub 2010 Oct 24. PMID 22432824